CLINICAL TRIAL: NCT05905497
Title: A Phase 1, Open-Label, Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Bemnifosbuvir in Healthy Adult Japanese Subjects
Brief Title: The Study of Bemnifosbuvir in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-018
Record Dates: First submitted 2023-04-20; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bemnifosbuvir (BEM) (Experimental): oral tablet
  Interventions: Drug: Bemnifosbuvir (BEM)

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM) — BEM administered BID for 4 days and QD on Day 5 (9 consecutive doses)
  Other Names: AT-527

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of Bemnifosbuvir in healthy adult Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/m2
* Willing to comply with the study requirements and to provide written informed consent
* The subject must have been born in Japan and have both parents and 4 grandparents of Japanese descent
* The subject must have lived outside of Japan for no more than 10 years

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of BEM Maximum plasma concentration (Cmax) | Day 1, Day 5
Pharmacokinetics (PK) of BEM Area under the plasma concentration-time curve (AUC) | Day 1, Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Cypress, California, United States